CLINICAL TRIAL: NCT05711862
Title: The Effects of Suvorexant on Sleep, Stress, and Cue-reactivity in Methamphetamine Use Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Heather E. Webber, PhD, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HSC-MS-22-0796
Record Dates: First submitted 2023-01-13; First posted 2023-02-03 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Methamphetamine Use Disorder
Keywords: sleeplessness; stress; Cue reactivity
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 week Placebo, then 1 week suvorexant (SUVO) (Experimental): After 1 week of placebo treatment there will be 1 week of wash out period before start of study medication
  Interventions: Drug: suvorexant (SUVO); Drug: Placebo
- 1 week suvorexant (SUVO), then 1 week Placebo (Experimental): After 1 week of SUVO treatment there will be 1 week of wash out period before start of placebo
  Interventions: Drug: suvorexant (SUVO); Drug: Placebo

INTERVENTIONS:
Drug: suvorexant (SUVO) — Participants will receive 20mg of SUVO for 7 days. Participants will be directed to take the medication between 9:30 PM and 10:00PM.
Drug: Placebo — Participants will receive 0mg of placebo for 7 days. Participants will be directed to take the medication between 9:30 PM and 10:00PM.

SUMMARY:
The purpose of this study is to determine the effects of SUVO on sleep, stress, and cue reactivity/craving and to evaluate the preliminary safety and side effects profile of suvorexant (SUVO)

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-5 criteria for MA use disorder
* Be fluent in English and able to understand the consent form

Exclusion Criteria:

* Have an alcohol use disorder or report binge drinking (>7 drinks for women and >14 drinks for men)
* Have a greater than mild substance use disorder on any other illicit substance
* Have any medical conditions contraindicating SUVO (e.g., severe pulmonary disease, severe cardiovascular disease or clinically abnormal ECG, severe liver or kidney disease, seizure disorder, or sleep disorder - particularly narcolepsy)
* Are currently taking medications with known drug interactions with SUVO (e.g., MAO inhibitors, anticonvulsants, haloperidol, phenothiazines, anesthetics, and any sedative)
* Are pregnant or breast feeding
* BMI > 30 (women only)
* Have a current DSM-5 psychiatric disorder or neurological disease requiring on-going treatment that would make participation unsafe
* Have history of seizure disorder
* Have a head injury with loss of consciousness in the last 5 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Webber, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 7 enrolled participants, 4 were randomized and 3 were lost to follow-up before randomization.
Period: First Intervention (1 Week)
Arm/Group | 1 Week Suvorexant (SUVO), Then 1 Week Placebo | 1 Week Placebo, Then 1 Week Suvorexant (SUVO)
Started | 2 | 2
Received Intervention | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Period: Washout (1 Week)
Arm/Group | 1 Week Suvorexant (SUVO), Then 1 Week Placebo | 1 Week Placebo, Then 1 Week Suvorexant (SUVO)
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | 1 Week Suvorexant (SUVO), Then 1 Week Placebo | 1 Week Placebo, Then 1 Week Suvorexant (SUVO)
Started | 2 | 1
Received Intervention | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes all participants who were randomized and received intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Week Suvorexant (SUVO), Then 1 Week Placebo | 1 Week Placebo, Then 1 Week Suvorexant (SUVO) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (5) | 38.5 (3.5) | 42.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4
Years of Education [Mean (Standard Deviation); unit: years] | 12 (1.4) | 13 (0) | 12.5 (1)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Sleep as Assessed by the PITTSBURGH SLEEP QUALITY INDEX (PSQI)
Description: Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21, higher score indicating a worse outcome. The global PSQI score is reported.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 1 Week SUVO: suvorexant (SUVO): Participants will receive 20mg of SUVO for 7 days in either the first the first or last week of the study. Participants will be directed to take the medication between 9:30 PM and 10:00PM.
- 1 Week Placebo: Placebo: Participants will receive 0mg of placebo for 7 days in either the first or last week of the study. Participants will be directed to take the medication between 9:30 PM and 10:00PM
Arm/Group | 1 Week SUVO | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
score on a scale | 8.66 (2.88) | 9.66 (0.57)

2. Primary Outcome: Resting State Alpha Power as Assessed by EEG
Description: EEG will be used to assess electrical activity in the brain, specifically, to assess alpha power, which is the level of activity in the 8-12Hz frequency range. Resting state EEG means that EEG will be assessed during wakeful rest. Alpha power will be assessed in each of the 4 brain lobes (frontal, central, parietal, and occipital) for 3 minutes during eyes closed wakeful rest and also for 3 minutes during eyes open wakeful rest. Alpha Power will be reported in microvolts squared (μV²). Higher alpha power indicates more sleepiness and lower alpha power indicates less sleepiness
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: microvolts squared (μV²)
Arm/Group | 1 Week SUVO | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
microvolts squared (μV²)
  Eyes closed - Fz (frontal) | -1.25 (0.25) | -1.12 (0.57)
  Eyes closed - Cz (Central) | -2.04 (0.52) | -1.42 (0.48)
  Eyes closed - Oz (occipital) | -1.19 (0.49) | -1.12 (0.75)
  Eyes closed - Pz (parietal) | -2.08 (0.27) | -1.78 (0.51)
  Eyes open - Fz (frontal) | -1.46 (0.21) | -1.25 (0.27)
  Eyes open - Cz (Central) | -2.16 (0.34) | -1.64 (0.44)
  Eyes open - Oz (occipital) | -1.55 (0.27) | -1.44 (0.71)
  Eyes open - Pz (parietal) | -2.36 (0.34) | -1.83 (0.34)

3. Primary Outcome: Amplitude of the Late Positive Potential (LPP) in Microvolts in Response to Visual Stimuli on the Picture Viewing Task as Assessed by the EEG
Description: The Picture Viewing Task will be used to elicit the late positive potential (LPP), reflecting the motivational salience of a stimulus. During this task, participants are asked to view a slideshow of images including pleasant, unpleasant, neutral, and Methamphetamine-related images. The amplitude of the LPP in microvolts in response to visual stimuli is reported.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | 1 Week SUVO | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
microvolts
  LPP Amplitude with Pleasant Images | 2.85 (0.96) | 1.60 (2.27)
  LPP Amplitude with Unpleasant Image | 1.90 (1.33) | 1.38 (1.37)
  LPP Amplitude with Methamphetamine Images | 1.62 (0.40) | 1.08 (0.27)
  LPP Amplitude with Neutral Images | 1.01 (0.85) | 0.67 (0.56)

4. Primary Outcome: Self-reported Stress as Assessed by the Stress Subscale of the Depression, Anxiety and Stress Scale (DASS-21)
Description: The Stress Subscale of the Depression, Anxiety and Stress scale (DASS-21) assesses stress levels. Total score on the DASS-21 stress subscale ranges from 0 to 21, with a higher score indicating greater stress.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 1 Week Suvorexant (SUVO): suvorexant (SUVO): Participants will receive 20mg of SUVO for 7 days in either the first the first or last week of the study. Participants will be directed to take the medication between 9:30 PM and 10:00PM.
Arm/Group | 1 Week Suvorexant (SUVO) | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
score on a scale | 7.67 (6.03) | 8.33 (8.50)

5. Primary Outcome: Self-reported Stress as Assessed by the Visual Analog Scale (VAS)
Description: The Visual Analog Scale is scored from 0-10, with 0 being no stress, 10 being extreme stress.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1 Week Suvorexant (SUVO) | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
score on a scale | 2.33 (3.21) | 5.67 (5.13)

6. Primary Outcome: Change of Cortisol Level
Description: During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. Saliva samples will be collected before and after the CPT, and cortisol levels in the saliva samples will be assessed. The change in cortisol level will be reported as [(cortisol level at post cold pressor task) - (cortisol level pre cold pressor task)].
Time Frame: baseline, about 32 minutes after the start of the cold pressor task
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | 1 Week SUVO | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
picograms per milliliter (pg/mL) | 2103.99 (4226.09) | 233.55 (1225.26)

7. Primary Outcome: Average Sleep Time Per Night Measured Nightly Via Actigraphy Watch Over 7 Nights
Description: The average sleep time per night (averaged over 7 days) will be reported.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: minutes per night
Arm/Group | 1 Week Suvorexant (SUVO) | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
minutes per night | 326.52 (113.90) | 303.14 (89.44)

8. Primary Outcome: Average Time Awake After Sleep Onset Measured Nightly Via Actigraphy Watch Over 7 Nights
Description: The average time awake after sleep onset per night (averaged over 7 days) will be reported.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: minutes per night
Arm/Group | 1 Week Suvorexant (SUVO) | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
minutes per night | 54.07 (20.13) | 44.89 (15.16)

9. Secondary Outcome: Number of Days of Methamphetamine Use as Assessed by the Time Line Follow Back (TLFB) Method
Description: Timeline Followback (TLFB) is a method to assess Methamphetamine use that involves asking study participants to self-report their Methamphetamine use over the past week.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 1 Week Suvorexant (SUVO) | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
days | 2.67 (2.52) | 3.33 (2.89)

10. Secondary Outcome: Number of Participants Positive for Methamphetamine Use as Assessed by the Urine Drug Screen (UDS)
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | 1 Week SUVO | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
Participants | 2 | 0

11. Secondary Outcome: Number of Participants Who Had Side Effects
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1 Week SUVO | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
Participants | 3 | 3

12. Secondary Outcome: Depression as Assessed by the Beck's Depression Inventory (BDI)Scale
Description: Beck's Depression Inventory (BDI)scale total score ranges from 0 to 63, higher score indicating more depression
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1 Week Suvorexant (SUVO) | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
score on a scale | 9.33 (3.06) | 25.00 (27.18)

13. Secondary Outcome: Suicidal Ideation and Behavior as Assessed by the COLUMBIA-SUICIDE SEVERITY RATING SCALE (CSSR)
Description: This is a semi-structured interview that measures suicide ideation on a 6-point ordinal scale, ranging from 0 (no suicide ideation) to 5 (suicidal intent with plan) with a higher score indicating worse outcome
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1 Week Suvorexant (SUVO) | 1 Week Placebo
Number analyzed (Participants) | 3 | 3
score on a scale | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: Up to 3 weeks
Description: Includes all participants who were randomized and received intervention.
Arm/Group | 1 Week Suvorexant (SUVO) | 1 Week Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Week Suvorexant (SUVO) (N=4) | 1 Week Placebo (N=4)
Drowsiness (Nervous system disorders) | 2 | 2
Not Sleeping Well (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 2 | 1
Nervousness (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 2
Sweating (Nervous system disorders) | 3 | 2
Cloudiness (Nervous system disorders) | 1 | 1
Memory Loss (Nervous system disorders) | 0 | 1
Fatigue Tiredness (Nervous system disorders) | 2 | 2
Difficulty Walking (Nervous system disorders) | 1 | 0
Weakness (Nervous system disorders) | 1 | 0
Heart Racing (Nervous system disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Stomach Cramps (Gastrointestinal disorders) | 0 | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Increased Urination (Renal and urinary disorders) | 2 | 0
Dry Mouth (General disorders) | 1 | 1
Fever or Chills (Immune system disorders) | 2 | 0
Muscle Aches (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT05711862/Prot_SAP_000.pdf